CLINICAL TRIAL: NCT03060655
Title: Randomized, Double Blind Trial of Study of PLGA-Mg Material in Clinical Orthopedics
Brief Title: Study of PLGA-Mg Material in Clinical Orthopedics
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYZ2017
Record Dates: First submitted 2017-01-18; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Fracture Dislocation
Keywords: PLGA-Mg; fracture; fixation; union
MeSH Terms: conditions — Fracture Dislocation; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLGA-Mg material (Placebo Comparator): The fixation of fragments of study group was accomplished with PLGA-Mg material.
  Interventions: Biological: PLGA-Mg material
- titanium alloy (Placebo Comparator): The fixation of fragments of control group was accomplished with titanium alloy material.
  Interventions: Biological: titanium alloy

INTERVENTIONS:
Biological: PLGA-Mg material — The PLGA-Mg material was used to accomplish the fixation of fragments. Then, the clinical outcome was assessed.
  Arms: PLGA-Mg material
Biological: titanium alloy — Traditional fixation was titanium alloy. the clinical outcome was assessed.
  Arms: titanium alloy

SUMMARY:
The different proportion samples of PLGA-Mg were made in this study. Then, they would be placed in the femoral condyle of the New Zealand rabbits. The appropriate proportion of PLGA-Mg is obtained after the experiment, which will be used to make the plate or screw to fix the fragments. Then, the clinical role for bone will be assessed.

DETAILED DESCRIPTION:
The deposition of calcium could be facilitated by the increase of magnesium, which played an important role in fracture union. However, its degradation may be completed before the fracture line was disappeared. In addition, the hydrogen may be released during degradation. Thus, its clinical popularization was limited.

As a new polymer material, poly lactic-co-glycolic acid (PLGA) has been widely used clinically. The hydrolytic production of PLGA was acidic, which could neutralize the alkalinity of production degraded from magnesium. In addition, it was a long time before the total accomplishment of degradation of PLGA, which may postpone the degradation of magnesium.

The different proportion samples of PLGA-Mg were made in this study. Their physical and chemical properties were analyzed to estimate its safety of implantation. Then, they would be placed in the femoral condyle of the New Zealand rabbits. The osteogenesis and complication of samples are examined to select an appropriate proportion of PLGA-Mg is obtained. Then, the PLGA-Mg material will be used to fix the fracture of human as a fixation. The review of the patients will be conducted to assess its clinical role.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Closed fracture
* Sign the agreement of the experiment

Exclusion Criteria:

* Pathologic fracture
* Open fracture
* Refused to participate
* Follow-up insufficient 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
fracture union time | 4 months

SECONDARY OUTCOMES:
complication | 1 months
  nonunion, toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ruipeng Zhang, M.D, Principal Investigator — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes